CLINICAL TRIAL: NCT02665728
Title: A Safety and Efficacy Evaluation of BLI400 Laxative in Constipated Adolescent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI400-201
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLI400 (Experimental): BLI400 Laxative
  Interventions: Drug: BLI400 Laxative

INTERVENTIONS:
Drug: BLI400 Laxative

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of BLI400 laxative in constipated adolescent subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at between 12-17 years of age
* Weight more than 40 kg (88 lbs.).
* Constipated, defined by the following criteria

  1. Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:

     1. Straining during > 25% of defecations
     2. Lumpy or hard stools in > 25% of defecations
     3. Sensation of incomplete evacuation for > 25% of defecations
  2. Loose stools are rarely present without the use of laxatives
  3. There are insufficient criteria for irritable bowel syndrome - loose (mushy) or watery stool in the absence of laxative use for more than 25% of bowel movements

Criteria A, B and C must be fulfilled for the last 12 weeks with symptom onset at least 6 months prior to diagnosis.

* Otherwise in good health, as determined by physical exam and medical history
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, intrauterine device, double-barrier method, depot contraceptive, sterilized, or abstinence)
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
* Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
* Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
* Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of Visit 3
* Subjects who are pregnant or lactating, or intend to become pregnant during the study
* Subjects of childbearing potential who refuse a pregnancy test
* Subjects who are allergic to the study medication
* Subjects taking narcotic analgesics or other medications known to cause constipation
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
* Subjects with an active history of drug or alcohol abuse
* Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
* Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (3):
- United States (3):
  - BLI Research Site 1, Miami, Florida
  - BLI Research Site 2, Palmetto Bay, Florida
  - BLI Research Site 3, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI400
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Arm/Group | BLI400
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Overall treatment response is defined as weekly response in at least 2 out of 4 weeks. Weekly response is defined as greater than or equal to 3 spontaneous bowel movements during a week.
Time Frame: 4 weeks
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | BLI400
Number analyzed (Participants) | 33
Participants | 32

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | BLI400
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 (N=33)
headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.